CLINICAL TRIAL: NCT05665023
Title: Single-arm Phase II Study of Bevacizumab Plus Modified FOLFIRINOX Chemotherapy in Ovarian, Fallopian Tube, or Primary Peritoneal Mucinous Carcinoma
Brief Title: Bevacizumab Plus Modiifed FOLFIRINOX in Ovarian, Fallopian Tube, or Primary Peritoneal Mucinous Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2021-1776
Record Dates: First submitted 2022-11-15; First posted 2022-12-27 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Mucinous Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: mucinous ovarian cancer; fallopian tube cancer; primary peritoneal cancer; palliative; avastin; modified FOLFIRINOX
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bevacizumab + modified FOLFIRINOX (Experimental): Bevacizumab 5mg/kg D1, oxaliplatin 85 mg/m2 D1 + leucovorin 400mg/m2 D1 + irinotecan 150 mg/m2 D1 + 5-FU 2,400 mg/m2 46h continuous infusion, every other week
  Interventions: Drug: Bevacizumab + modified FOLFIRINOX

INTERVENTIONS:
Drug: Bevacizumab + modified FOLFIRINOX — Bevacizumab 5mg/kg D1, oxaliplatin 85 mg/m2 D1 + leucovorin 400mg/m2 D1 + irinotecan 150 mg/m2 D1 + 5-FU 2,400 mg/m2 46h continuous infusion, every other week

SUMMARY:
This research study is evaluating a modified FOLFIRINOX plus bevacizumab therapy for mucinous ovarian cancer, fallopian tube cancer, and primary peritoneal cancer.

DETAILED DESCRIPTION:
This study is aimed at recurrent/metastatic/resectable patients who have received systemic chemotherapy of 2nd line or less. Excludes previously diagnosed mucinous tumors of gastrointestinal origin through upper and lower endoscopy and pathologic immunohistochemical staining.

Bevacizumab plus modified FOLFIRINOX drug is administered every 2 weeks. To prevent neutropenia fever during chemotherapy, pegteograstim is given 24 hours after chemotherapy.

The primary objective of this study is the objective response rate (ORR). The secondary objectives are progression-free survival (PFS) and disease control rate at 6 months after administration, disease control rate (DCR), overall survival (OS), drug safety, and quality of life improvement as assessed by patient questionnaires.

In addition, the investigators intend to explore biomarkers that can predict the effect of bevacizumab + mFOLFIRINOX combination therapy through the collection of tumor samples and blood samples for exploratory purposes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recurrent, metastatic, or unresectable ovarian cancer, fallopian tube cancer, or primary peritoneal cancer diagnosed cytologically or histologically as mucinous cancer.

   *Subjects who are metastatic (stage IV) or mucinous ovarian cancer that cannot be surgically resected at diagnosis may have undergone cytoreductive surgery prior to systemic chemotherapy. It is appropriate for participation in this study if there are residual lesions after surgery and other selection criteria are met.
2. Mucous tumors of gastrointestinal origin should be excluded by prior upper and lower intestinal endoscopy and pathologic immunohistochemical staining (CEA, SATB2, etc.).
3. Patients who have not received previous systemic chemotherapy for recurrent, metastatic, or unresectable ovarian, fallopian tube, or primary peritoneal cancer, or who have failed second-line or less systemic chemotherapy. However, immunotherapy alone (eg, anti-PD-1 or anti-PD-L1 immunotherapy) is not included in previous chemotherapy.

   *Platinum susceptibility does not affect the selection/exclusion criteria for this trial.
4. Informed consent
5. Age more than 19 years old
6. Patients with measurable lesions according to RECIST v1.1.
7. ECOG Performance score 0-2
8. Patients with adequate organ function
9. Women of childbearing potential must either have a negative pregnancy test on a urine or serological test or consent to the use of an appropriate contraceptive method.

Exclusion Criteria:

1. Patients who have previously received systemic chemotherapy, including oxaliplatin or irinotecan. *Previous treatment with bevacizumab is acceptable.
2. Pregnant or breastfeeding women
3. Patients who received chemotherapy, targeted small-molecule agents, or radiotherapy within 2 weeks prior to Day 1 of the study, or who have not yet recovered (Grade 1 or lower or baseline level) from a previously administered drug-induced adverse event.
4. Active central nervous system (CNS) metastases and/or carcinoma meningitis.
5. Patients with known aggravation within the past 3 years or other malignant tumors requiring aggressive treatment.
6. Patients with moderate acute or chronic medical conditions or abnormal findings on examination, which are judged to affect the results of this study
7. Infected with Human Immunodeficiency Virus (HIV) (HIV-1/2 antibody) infection or active hepatitis B (HBsAg positive and HBV DNA ≥100 copies/ml) or hepatitis C (anti-HCV antibody positive and HCV RNA detected) being)
8. Clinically significant heart disease.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2022-10-28 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | up to 1 year
  Objective response rate assessed using Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1) for Intention-to-treatment group

SECONDARY OUTCOMES:
Progression-free survival | up to 1 year
  Progression-free survival assessed using Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1) and Kaplan-Meier Survival analysis
Disease control rate | at 6 months
  Disease control rate assessed using Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1) for Intention-to-treatment group
Overall survival | up to 1 year
  Overall survival assessed using Kaplan-Meier Survival analysis to check survival outcomes of Intention-to-treatment group
Number of Participants With Adverse Events (CTCAE v5.0) | from the start to within 30 days of the final chemotherapy
  Safety profiles assessed using Common Terminology Criteria for Adverse Events v5.0 (CTCAE v5.0)
Patient reported outcomes | at the beginning and every 4 cycles of the treatment (each cycle is 14 days), up to 1 year
  Patient reported outcomes assessed using EQ-5D
Patient reported outcomes | at the beginning and every 4 cycles of the treatment (each cycle is 14 days), up to 1 year
  Patient reported outcomes assessed using EORTC QLQ-CIPN20
Febrile neutropenia prevention efficacy and safety profiles of Pegteograstim | from the start to within 30 days of the final chemotherapy
  Pegteograstim efficacy and safety profiles assessed using Common Terminology Criteria for Adverse Events v5.0 (CTCAE v5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Min Hwan Kim, Principal Investigator — Division of Medical Oncology, Yonsei Cancer Center, Yonsei Univ. College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No